CLINICAL TRIAL: NCT07041970
Title: PregFit Adventure: Strengthening Mothers-to-Be
Brief Title: PregFit Adventure: Strengthening Mothers-to-Be (PregFit)
Acronym: PregFit
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Sergio Martínez Vázquez, Doctor, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PregFit-Jun-25
Record Dates: First submitted 2025-06-16; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Pregnant Women; Exercise; Game
Keywords: pregnant women; exercise; physical condition; exergames; low-risk pregnancy; physical activity
MeSH Terms: conditions — Motor Activity | interventions — Exergaming

STUDY DESIGN:
Intervention Model Description: * Intervention Group: The program consists of using the device, a minimum of 30 minutes per session two to three times per week and not exceeding ≥3 hours, for at least 8 weeks up to a maximum of 3 months or until the onset of discomfort disabling physical activity, with the minimum time for intervention being at least 8 weeks. Exercise based on exergames will be performed including at least 10 minutes of warm-up and 10 minutes of cool-down, and under the supervision of a licensed health professional.
  * Control Group: Low-risk pregnant women who have normal pregnancy follow-up with Health Education received in childbirth preparation classes and maternal education received in routine pregnancy care by primary and specialized care midwives.
Who Masked: Outcomes Assessor
Masking Description: Masking: Unique (Results Evaluator).
  Description of masking: Due to the design of the study and the nature of the interventions, it is impossible to mask staff and participants at the care centers. The evaluators, who measure the outcomes, and the interpreter, who analyzes the data, will be masked in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): @Intervention Group: The program consists of using the device, a minimum of 30 minutes per session two to three times per week and not exceeding ≥3 hours, for at least 8 weeks up to a maximum of 3 months or until the onset of discomfort disabling physical activity, with the minimum time for intervention being at least 8 weeks. Exercise based on exergames will be performed including at least 10 minutes of warm-up and 10 minutes of cool-down, and under the supervision of a licensed health professional.
  Interventions: Other: Exergame
- Control (No Intervention): @Control Group: Low-risk pregnant women who have normal pregnancy follow-up with Health Education received in childbirth preparation classes and maternal education received in routine pregnancy care by primary and specialized care midwives.

INTERVENTIONS:
Other: Exergame — The training program will focus on strength and functional movements. It requires a Nintendo Switch console, a Ring-Con (a Pilates ring that the user holds or ring holder), wireless Joy-Con controllers (the right Joy-Con, connected to the Ring-Con; and the left Joy-Con, attached to the strap around the player's thigh) and a screen. In adventure mode, women will move through the game by performing physical activities such as jogging or doing squats. To minimize risk, knee-assist mode will be used, which makes the game more accessible. Activating knee assist mode provides support when women perform exercises that require walking, kneeling or squatting, making these activities easier for pregnant women, increasing the fitness benefits of the game. In battle mode women will perform aerobic activities, strength training and yoga exercises that involve the whole body to advance in the game.
  Arms: Intervention

SUMMARY:
1. Design.

   This will be a randomized clinical trial (RCT) with two groups, an experimental or intervention group and a control group.
2. Population, criteria, sample, calculation.

   The study population will be low-risk pregnant women.

   Inclusion criteria:
   * Pregnant women at low obstetric risk and with no musculoskeletal or health problems affecting their physical condition, ability to exercise or participate in the exergame activities.
   * Read the information sheet and sign the informed consent form to agree to take part in the study.
   * >18 years of age
   * Spanish comprehension and communication skills
   * Able to perform physical activity related to the use of the device for at least 30 minutes, 2-3 times a week, for at least 8 weeks

   Exclusion criteria:
   * Failure to meet any of the inclusion criteria
   * Giving birth during the procedure and at least 8 weeks of device use have not elapsed.

   Assignment: All women receiving maternal education from all participating health centers will be randomized to ensure that there is no sample contamination and their relevance to the intervention or control group will be established according to randomization.

   Sample size calculation: It was estimated that the number of participants should be at least 15% for this pilot study of what would be a future intervention project. Using self-perceived physical fitness as the dependent variable, and in validation studies having had samples of around 160 women (Romero-Gallardo et al., 2020), at least 24 women will be needed in the single intervention group for this pilot study. Similarly, at least 24 women in the control group are needed for comparison. It is estimated that 20% of women may drop out of the intervention before the minimum 8 weeks, thus establishing a sample size of at least 30 women to recruit. Using similar studies (Tuan et al., 2024) as a reference, we will try to reach the ideal sample size of 42 healthy pregnant women who complete the intervention and at least 42 for the control group who receive routine pregnancy follow-up EpS and antenatal classes.
3. Description of the intervention.

   * Intervention Group: The program consists of using the device, a minimum of 30 minutes per session two to three times per week and not exceeding ≥3 hours, for at least 8 weeks up to a maximum of 3 months or until the onset of discomfort disabling physical activity, with the minimum time for intervention being at least 8 weeks. Exercise based on exergames will be performed including at least 10 minutes of warm-up and 10 minutes of cool-down, and under the supervision of a licensed health professional.

The training program will focus on strength and functional movements. It requires a Nintendo Switch console, a Ring-Con (a Pilates ring that the user holds or ring holder), wireless Joy-Con controllers (the right Joy-Con, connected to the Ring-Con; and the left Joy-Con, attached to the strap around the player's thigh) and a screen. In adventure mode, women will move through the game by performing physical activities such as jogging or doing squats. To minimize risk, knee-assist mode will be used, which makes the game more accessible. Activating knee assist mode provides support when women perform exercises that require walking, kneeling or squatting, making these activities easier for pregnant women, increasing the fitness benefits of the game. In battle mode women will perform aerobic activities, strength training and yoga exercises that involve the whole body to advance in the game. Women will receive in-game coin rewards, character customization and level progression based on exercise volume, which encourages improvement of their skills. As an example, with the assisted knee mode, women will have to squeeze and stretch the titular ring working muscles such as the trapezius, triceps, pectoralis major and minor and abdominal muscles. In addition, to go about defeating the monsters they will have to do shoulder abduction and adduction exercises, internal and external rotation of the shoulders and flexion of the elbow as shown in the images of the orientation trailer, provided to women and available in this memory.

@Control Group: Low-risk pregnant women who have normal pregnancy follow-up with Health Education received in childbirth preparation classes and maternal education received in routine pregnancy care by primary and specialized care midwives.

Masking: Unique (Results Evaluator).

Description of masking: Due to the design of the study and the nature of the interventions, it is impossible to mask staff and participants at the care centers. The evaluators, who measure the outcomes, and the interpreter, who analyzes the data, will be masked in this study.

Place: It will take place in a health center, which is part of the ecosystem of the Andalusian Health Service.

DETAILED DESCRIPTION:
1. PROJECT DATA

   PI (Name and surname): Martínez Vázquez, Sergio; svazquez@ujaen.es; Tel: +34 953212014

   PregFit Adventure: Strengthening Mothers-to-Be
2. SCIENTIFIC EXCELLENCE, NOVELTY AND RELEVANCE OF THE PROPOSAL.

   It is estimated that up to 5 million deaths per year could be avoided if the world's population were more physically active. Therefore, the World Health Organization (WHO) promulgates guidelines on physical activity and sedentary lifestyles, emphasizing that all people, regardless of age or ability, can be active and that any movement counts. Physical activity, is defined as any bodily movement produced by the contraction of skeletal muscles. Exercise, on the other hand, is defined as physical activity consisting of planned, structured, repetitive body movements performed to improve one or more components of physical fitness. It is an essential element that is part of a healthy lifestyle, and obstetrics-gynecology professionals as well as other obstetric care professionals should encourage women to continue or begin exercising as an important component of optimal health.

   There are recommendations for at least 150 minutes of moderate-intensity aerobic activity per week during pregnancy and postpartum. The guidelines recommend that women who routinely engaged in vigorous-intensity aerobic activity or who were physically active before pregnancy can continue these activities during pregnancy and postpartum. In addition, pregnant women should be under the care of an obstetrics-gynecology professional who can monitor the progress of the pregnancy.

   Physical inactivity is the fourth leading risk factor for early mortality worldwide. During pregnancy, physical inactivity and excessive weight gain have been recognized as independent risk factors for maternal obesity and pregnancy-related complications, including gestational diabetes mellitus (GDM). It also reduces the risk of excessive gestational weight gain, gestational hypertensive disorders, low birth weight, preterm delivery, or cesarean section.

   There is no evidence that regular physical activity during pregnancy can cause miscarriage, poor fetal growth, musculoskeletal injury, or preterm delivery in women with uncomplicated pregnancies. In addition, regular physical activity has been associated with an increased likelihood of having a vaginal delivery. In the absence of obstetric and medical complications or contraindications, physical activity during pregnancy is safe and desirable, and pregnant women should be encouraged to continue or initiate safe physical activities. Some of these activities defined as safe include: walking, stationary cycling, aerobic exercise, dancing, resistance exercises (e.g., weights, elastic bands), stretching exercises, hydrotherapy, or water aerobics.

   Ring Fit Adventure is an interactive exercise game for the Nintendo Switch console that combines physical activity with elements of play and fun. The game involves stretching movements, balance, and moderate aerobic exercise, which can be beneficial if performed properly. The intensity of the exercise can vary and it is important for pregnant women to adjust their effort so as not to overtax their bodies. It defeats monsters through exercise, shoulder presses, or yoga poses. It has a holder ring, this is a control device that is used for resistance exercises, and there is also a leg strap that tracks running pace. The game is not specifically designed for pregnant women, and some movements, such as jumping or performing certain quick stretches, may not be appropriate during advanced pregnancy, although, when starting, the game performs some tests to gauge strength, running speed, and intensity level. In addition, it has an "assisted mode," which allows adjustments for shoulder accessibility, knee assistance, back assistance, or ab assistance. For example, instead of doing a squat or ring squeeze, a button is pressed or cool-down periods are given for repeat attacks allowing the woman to rest.

   Nintendo Ring Fit Adventure, considered an "exergame" or games that encourage exercise while playing, has been shown to be effective in older adult populations by significantly improving muscle mass, strength and functionality or reducing falls in different clinical trials. The results are also very positive if the study population had musculoskeletal problems, osteoarthritis or chronic low back pain. Benefits related to weight loss in overweight and obese patients have also been described.

   However, there are hardly any studies carried out in pregnant women that propose physical exercise interventions and then evaluate the effect that these interventions have on their physical condition or level of physical activity. Moreover, the few studies that contemplate this type of approach use recommendations and physical exercise guidelines that do not take into account new technologies or immersive gamification, such as exergames. Therefore, the objective is to evaluate an exergame-based exercise training program administered through Nintendo Ring Fit Adventure and to study its effect on the physical condition of pregnant women and their level of activity.
3. RESEARCH TEAM

Sergio Martínez Vázquez (IP) (SMV) - Professor - University of Jaén

4. OBJECTIVES AND HYPOTHESES

Hypothesis: After participating in the Exergame-based training program using Ring Fit Adventure, pregnant women will improve their self-perceived physical fitness and physical activity level, showing a statistically significant increase in both indices.

General Objective: To evaluate an exergame-based exercise training program administered through Nintendo Ring Fit Adventure and to study its effect on the fitness and physical activity level of pregnant women.

In order to achieve the general objective, the following specific objectives are set:

1. Determine the physical condition and physical activity level of pregnant women prior to training.
2. To determine the physical condition and physical activity level of pregnant women after training.

5. METHODOLOGY

1. Design.

   This will be a randomized clinical trial (RCT) with two groups, an experimental or intervention group and a control group.
2. Population, criteria, sample, calculation.

   The study population will be low-risk pregnant women.

   Inclusion criteria:

   • Pregnant women at low obstetric risk and with no musculoskeletal or health problems affecting their physical condition, ability to exercise or participate in the exergame activities.

   • Read the information sheet and sign the informed consent form to agree to take part in the study.
   * >18 years of age
   * Spanish comprehension and communication skills
   * Able to perform physical activity related to the use of the device for at least 30 minutes, 2-3 times a week, for at least 8 weeks

   Exclusion criteria:

   • Failure to meet any of the inclusion criteria

   • Giving birth during the procedure and at least 8 weeks of device use have not elapsed.

   Assignment: All women receiving maternal education from all participating health centers will be randomized to ensure that there is no sample contamination and their relevance to the intervention or control group will be established according to randomization.

   Sample size calculation: It was estimated that the number of participants should be at least 15% for this pilot study of what would be a future intervention project. Using self-perceived physical fitness as the dependent variable, and in validation studies having had samples of around 160 women, at least 24 women will be needed in the single intervention group for this pilot study. Similarly, at least 24 women in the control group are needed for comparison. It is estimated that 20% of women may drop out of the intervention before the minimum 8 weeks, thus establishing a sample size of at least 30 women to recruit. Using similar studies as a reference, we will try to reach the ideal sample size of 42 healthy pregnant women who complete the intervention and at least 42 for the control group who receive routine pregnancy follow-up EpS and antenatal classes.
3. Description of the intervention.

   @Intervention Group: The program consists of using the device, a minimum of 30 minutes per session two to three times per week and not exceeding ≥3 hours, for at least 8 weeks up to a maximum of 3 months or until the onset of discomfort disabling physical activity, with the minimum time for intervention being at least 8 weeks. Exercise based on exergames will be performed including at least 10 minutes of warm-up and 10 minutes of cool-down, and under the supervision of a licensed health professional.

   The training program will focus on strength and functional movements. It requires a Nintendo Switch console, a Ring-Con (a Pilates ring that the user holds or ring holder), wireless Joy-Con controllers (the right Joy-Con, connected to the Ring-Con; and the left Joy-Con, attached to the strap around the player's thigh) and a screen. In adventure mode, women will move through the game by performing physical activities such as jogging or doing squats. To minimize risk, knee-assist mode will be used, which makes the game more accessible. Activating knee assist mode provides support when women perform exercises that require walking, kneeling or squatting, making these activities easier for pregnant women, increasing the fitness benefits of the game. In battle mode women will perform aerobic activities, strength training and yoga exercises that involve the whole body to advance in the game. Women will receive in-game coin rewards, character customization and level progression based on exercise volume, which encourages improvement of their skills. As an example, with the assisted knee mode, women will have to squeeze and stretch the titular ring working muscles such as the trapezius, triceps, pectoralis major and minor and abdominal muscles. In addition, to go about defeating the monsters they will have to do shoulder abduction and adduction exercises, internal and external rotation of the shoulders and flexion of the elbow as shown in the images of the orientation trailer, provided to women and available in this memory.

   @Control Group: Low-risk pregnant women who have normal pregnancy follow-up with Health Education received in childbirth preparation classes and maternal education received in routine pregnancy care by primary and specialized care midwives.

   Masking: Unique (Results Evaluator).

   Description of masking: Due to the design of the study and the nature of the interventions, it is impossible to mask staff and participants at the care centers. The evaluators, who measure the outcomes, and the interpreter, who analyzes the data, will be masked in this study.

   Place: It will take place in a health center, which is part of the ecosystem of the Andalusian Health Service, having HD TV with HDMI connection to support the device, as well as good conditions of space, lighting and habitability that favor the comfort of the participating pregnant women. This will be detailed in the request for permission to the CEIH of the province of Jaén, requesting authorization from the center.
4. Recruitment and follow-up.

   Women will be recruited at their first contact with pregnancy care and follow-up care, whether in primary or specialized care, through the midwives who provide this care in the aforementioned units.
5. Sources of information and target variables of the study.

   In the first phase, women will be recruited who, after learning about the objectives of the project, voluntarily decide to participate. All of them will answer a self-administered questionnaire that will include sociodemographic variables, obstetric history and physical exercise before and during pregnancy, using the short version of the International Physical Activity Questionnaire (IPAQ) (IPAQ-SF), which quantifies physical activity during the last seven days, divided into four categories: vigorous intensity, moderate intensity, walking and sitting. In addition to intensity, the frequency and duration of physical activity are assessed. It includes 7 items on the "last 7 days" with items such as "During the last 7 days, how many days did you perform vigorous physical activities such as heavy lifting, digging, aerobic exercise, running or cycling at high speed?", with responses from 0 to 7. The response categories are divided into "don't know", "10 min", "20 min", and so on up to "2 h or more". The tool is validated in pregnant women which allows assessing the level of physical activity in this population, including the frequency, duration and intensity of the activity performed.

   It will also include the International Fitness Scale-IFIS, previously validated in the Spanish pregnant population. It is an assessment tool designed to measure adults' perception of their general fitness status. It was developed in order to provide a simple and quick way to obtain information on different dimensions of physical fitness, without the need for complex physical tests, assessing: Aerobic capacity or cardiovascular endurance, muscular strength, muscular endurance, flexibility, speed and agility. The answers are given on a Likert scale of 5 options: Very bad, Bad, Acceptable, Good and Very good. The higher the score, the better the self-perception of general physical fitness. It has been adapted to different populations and sociocultural contexts.

   For the inclusion criteria, low-risk pregnant women of legal age, with no incapacity to understand Spanish, of any week of gestation up to the moment of delivery will be selected, provided that the woman had no discomfort to perform the physical activity. Women with risky pregnancies or any health condition or pathology that makes physical exercise difficult will be excluded. Then, once the sample is known, the program guidelines will be designed in a second phase. For the determination of the training program guidelines, the recommendations of various public entities such as the American College of Gynaecologyst (ACOG), U.S. Department of Health and Human Services as well as references from other studies conducted in sociocultural contexts similar to the study population will be followed. These recommendations indicate that it should be at least 150 minutes of moderate-intensity aerobic activity per week during pregnancy , distributed throughout the week, establishing a minimum device use of 30 minutes per session two to three times per week and not exceeding ≥3 hours per week of use.

   In the next phase, all women will be advised to attend the study center at least 2 to 3 times a week, for the duration of gestation or until the onset of discomfort that disables physical activity, with the minimum time for the intervention being 8 weeks to 3 months, due to the positive results associated with this duration in similar studies in other populations. Before starting the use of the device, a first session will be held to explain its use to the pregnant women, as well as to provide them with a self-explanatory trailer available on the YouTube platform (https://www.youtube.com/watch?v=RvaJJIRIBt8&t=58s).

   In the last phase, the questionnaire will be administered again to the participants when at least 8 weeks, and up to three months, have elapsed since the beginning of the intervention or delivery has occurred in that time frame, answering the questionnaire without taking into account the time of delivery, and not considering the delivery situation.
6. Analysis.

   The statistical program used for data analysis will be SPSS 28.0. First, descriptive statistics will be determined using absolute and relative frequencies for categorical variables and means with standard deviations for quantitative variables. Preliminary checks will be carried out to analyze the normality of the data and homoscedasticity. To compare demographic data between the intervention and control groups, appropriate statistical tests including the chi-square, 2-tailed t-test and Mann-Whitney U test will be used depending on the data and their distribution characteristics. To address potential attrition, an intention-to-treat (ITA) analysis, which incorporates a simple imputation technique, will be used. Specifically, for missing data, the last observation carried forward method will be used. To assess the effects of the intervention on outcomes over time, a mixed ANOVA will be used, designating time as the within-participant variable and the nature of the intervention as the between-participant variable. For any significant interaction or main effect, post hoc assessments were performed using the Bonferroni test.
7. Limitations and contingency plan.

Selection bias due to non-representative participation of the study population. In this sense, comparisons will be made to see the similarities with the reference population in terms of variables such as age, level of education, etc. Confounding bias due to the nature of the study, although it will be considered, the researchers don´t believe that its influence will be differential. This is intended to be controlled both from the design with the selection of the study subjects with adequate inclusion and exclusion criteria; subsequently with the data analysis, adjusting the multivariate analysis for all those variables that could confound the results. However, due to the timing of the data collection, is not believed that this problem will occur, since the women will be given precise instructions on how to answer the questionnaire and will be given a contact telephone number and e-mail to resolve any doubts they may have. There may be some variability with respect to the intervention, since some women can carry it out for 8 weeks and others for 3 months, depending on the duration of their pregnancy, although considering that the sample of pregnant women, despite being low risk, may have different weeks of gestation and different delivery dates from the time of recruitment, this has been taken into account in the design of the temporality of the intervention, establishing time limits in accordance with the results demonstrated in the evidence in similar studies. The main strength of the study is its novelty and originality, given that there are no studies on this subject in the Spanish context. Another strength is the experience of the research team in working with the study population, being a mixed, multidisciplinary group of researchers with a large representation of midwives.

6. ETHICAL CONSIDERATIONS

The research protocol has been registered in Clinical Trials (https://clinicaltrials.gov/) with the code: XXXXX. All participants will be asked for informed consent in accordance with Law 14/2007, of 3 July, on Biomedical Research and at all times the Organic Law 3/2018, of 5 December, on the Protection of Personal Data and Guarantee of Digital Rights will be applied. To guarantee said informed consent, an information sheet will be given to each woman prior to her participation. Approval is requested from the Research Ethics Committee of Jaén (CEI/CEIM Provincial de Jaén).

7. CHRONOGRAM AND DISTRIBUTION OF TASKS

1 2 3 4 5 6 7 8 9 10 11 12 2025 1 1 2 2 2 2026 1 2 3 4 5 6 7 8 9 10 11 12 3 3 3 3 3 3 3 3 3 3 4 4

Distribution of phases throughout the project execution period.

8. TRANSFER PLAN

The results and analysis obtained will be transferred to;

1. Federation of Spanish Midwives Associations (FAME), Society of Obstetrics and Gynecology (SEGO).
2. TTOs and similar units for the management and evaluation of the transfer in R&D centers.
3. National civilian agencies for pregnancy, childbirth and puerperium.
4. Andalusian Health Service (SAS).

The results obtained will be used for the development of a clinical practice guideline (CPG) on safe physical activity during pregnancy. The training derived from the clinical practice guidelines will also empower healthcare professionals to better care for pregnant women.

9. REQUESTED BUDGET

Personnel costs: Tasks will be distributed among the members of the research team and no hiring of personnel will be necessary - 0 Inventory costs: Ring Fit Adventure - 69,99€. Nintendo Switch 2 - 469,99€. Space costs: Available and conditioned space in the health center will be used - 0€.

Publication costs: we estimate an average open cost of USD 3630 (approx. 3176.41 €), taking Midwifery magazine as an example, since it is a reference in its field.

Total budgeted: 69.99 + 469.99 + 3176.41 (x21% Indirect costs) = 3716.39 (21%) = 4497.

10. EXPECTED RESULTS

Improved physical fitness and physical activity of low-risk pregnant women participating in the intervention:

* Significant improvements in physical condition parameters.
* Increase in the level of habitual physical activity.
* Potential reduction of discomfort and improvement in psychological state.

Moreover, it lies in its importance:

* To demonstrate that exergames can be an effective, safe and motivating tool to promote physical activity in pregnant women.
* Contribute to the formulation of recommendations and health programs that integrate innovative technology in prenatal care.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women at low obstetric risk and with no musculoskeletal or health problems affecting their physical condition, ability to exercise or participate in the exergame activities.
* Read the information sheet and sign the informed consent form to agree to take part in the study.
* >18 years of age
* Spanish comprehension and communication skills
* Able to perform physical activity related to the use of the device for at least 30 minutes, 2-3 times a week, for at least 8 weeks

Exclusion Criteria:

* Failure to meet any of the inclusion criteria
* Giving birth during the procedure and at least 8 weeks of device use have not elapsed.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women (cis).
Enrollment: 84 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-12-26 (Estimated); Study Completion 2026-12-26 (Estimated)

PRIMARY OUTCOMES:
Increase in the level of habitual physical activity - Short version of the International Physical Activity Questionnaire (IPAQ-SF) | From 8 weeks to 3 months
  Short version of the International Physical Activity Questionnaire (IPAQ) (IPAQ-SF), which quantifies physical activity during the last seven days, divided into four categories: vigorous intensity, moderate intensity, walking and sitting. In addition to intensity, the frequency and duration of physical activity are assessed. It includes 7 items on the "last 7 days" with items such as "During the last 7 days, how many days did you perform vigorous physical activities such as heavy lifting, digging, aerobic exercise, running or cycling at high speed?", with responses from 0 to 7. The response categories are divided into "don't know", "10 min", "20 min", and so on up to "2 h or more". The tool is validated in pregnant women which allows assessing the level of physical activity in this population, including the frequency, duration and intensity of the activity performed.
Significant improvements in physical condition parameters - International Fitness Scale-IFIS | From 8 weeks to 3 months.
  The International Fitness Scale-IFIS, previously validated in the Spanish pregnant population. It is an assessment tool designed to measure adults' perception of their general fitness status. It was developed in order to provide a simple and quick way to obtain information on different dimensions of physical fitness, without the need for complex physical tests, assessing: Aerobic capacity or cardiovascular endurance, muscular strength, muscular endurance, flexibility, speed and agility. The answers are given on a Likert scale of 5 options: Very bad, Bad, Acceptable, Good and Very good. The higher the score, the better the self-perception of general physical fitness. It has been adapted to different populations and sociocultural contexts.

IPD SHARING:
Plan to Share IPD: Undecided